CLINICAL TRIAL: NCT04879186
Title: A Retrospective Cohort Study Investigating the Risk Factors and Long-term Outcome of Contrast Induced Nephropathy Among Vascular Patients Undergoing Lower Limb Angioplasty
Brief Title: Contrast Induced Nephropathy Among Vascular Patients Undergoing Lower Limb Angioplasty
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2020/2659
Record Dates: First submitted 2021-05-04; First posted 2021-05-10 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Contrast-induced Nephropathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing peripheral endovascular angioplasty: Patients undergoing peripheral endovascular angioplasty. No intervention other than what was already completed as part of routine clinical care, as this is a retrospective cohort.
  Interventions: Procedure: Peripheral endovascular angioplasty

INTERVENTIONS:
Procedure: Peripheral endovascular angioplasty — Peripheral endovascular angioplasty - using endovascular techniques to treat peripheral artery occlusive lesions.

SUMMARY:
Contrast induced nephropathy (CIN) is an iatrogenic renal injury following intravascular administration of radio-opaque contrast media (CM) in susceptible individuals. As the third leading cause of hospital acquired renal failure, it is associated with increased mortality, morbidity and prolonged hospital stay. Endovascular procedures have gained greater popularity in the past decade due to the advance in technology. This has also led to the increased incidence of CIN after vascular surgeries. We are conducting a retrospective cohort study in Singapore General Hospital using our perioperative database collected in the past five years.

We will be extracting relevant patient perioperative information including both clinical diagnosis and lab values. Our primary aim is to establish the incidence of CIN among vascular patients with or without pre-existing chronic renal impairment undergoing elective peripheral endovascular angioplasty. Our secondary aims are to establish the risk factors and protective factors that lead to the development of CIN in vascular patients after peripheral endovascular angioplasty. We will also be looking at the long-term outcome of patients who have developed CIN after vascular endovascular angioplasty. The results of the study will enable us to identify patients at high risk of development of CIN, thus appropriate measures can be initiated early and help with their recovery process.

DETAILED DESCRIPTION:
We propose a retrospective single-center cohort study conducted in Singapore general hospital. Data would be extracted in patients who have undergone peripheral endovascular angioplasty from 01/01/2015 to 01/01/2020. The data will be extracted from the eHINTs Perioperative Subject Area without any direct identifiers. The subject area has been previously curated as part of the SingHealth ODySSEy (On-prem Research Data Science and Systems Explorer) System. There will be no patient identifier collected and the data collection administration will not have any access to patient identifier. Waiver of consent is sought and no patient interaction would be required for the study.

The parameters to be extracted would include preoperative data such as patient demographics (age, gender, race, BMI), baseline comorbidities including but not limited to: hypertension, hyperlipidemia, diabetes mellitus, smoking, anemia, heart diseases (previous heart attack/history of congestive heart failure), preoperative renal function (measured by baseline Urea, creatinine, electrolytes level Na, K, Cl), preoperative long-term medication use including ACE inhibitor, ARB, beta-blocker, statin and diuretics and NSAIDS. Intraoperative data including types of anaesthesia used, operative duration, presence of intraoperative hypotension. Postoperative parameters such as mortality, length of stay in hospital and ICU, postoperative renal function measured by urea and creatinine level within 3 days and one month postoperatively.

Statistical analysis will be performed to study the risk factors for CIN in patients undergoing peripheral endovascular angioplasty.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing peripheral endovascular angioplasty during the study period, at Singapore General Hospital

Exclusion Criteria:

* Patients < 21 years of age

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient data is drawn from the eHINTs Perioperative Subject Area, a previously curated datat mart which forms part of the SingHealth ODySSEy (On-prem Research Data Science and Systems Explorer) System. This is a registry of all patients who have undergone surgery in Singapore General Hospital. Patient identifier are removed before data release to the study team.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2015-07-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Contrast induced nephropathy | 1 week post procedure
  Rise in creatinine post operatively according to KDIGO criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
No current plan, as a fresh application is needed for each access to data.